CLINICAL TRIAL: NCT03373448
Title: Treatment of Mild to Moderate Peri-implantitis Using an Oscillating Chitosan Device Versus Titanium Curettes - a Multicenter Randomized Clinical Trial
Brief Title: Treatment of Mild to Moderate Peri-implantitis Using an Oscillating Chitosan Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Labrida AS (Industry)
Responsible Party: Principal Investigator, Caspar Wohlfahrt, Specialist i periodontology, Labrida AS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 256756
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Patients will be allocated either to test (Labrida BioClean® or control (titanium curettes) treatment by computer-generated block randomization to ensure equal sample sizes. The examiners will be blinded to the treatment allocation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Examiners blinded to treatment allocation since treatment is performed by a dental hygienist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labrida BioClean (Active Comparator): Labrida BioClean- chitosan device.The brush bristles of the test device (Labrida BioClean® LABRIDA AS, Oslo Norway) are made of the biopolymer chitosan. Any debris left from the chitosan bristles is completely biocompatible and will dissolve or be resorbed thus not causing harm to the tissues surrounding the implant. Chitosan is made from chitin derived from shell of marine crustaceans such as shrimp and crab, however chemically modified and thus not even considered to be animally derived. Chitosan has been approved for use in e.g., surgical bandages, as a haemostatic agent and as dietary supplement used in a wide range of nutritional and health products. Chitosan has also been documented to be non-allergenic and it has been suggested that chitosan has anti-inflammatory properties.
  Interventions: Device: Labrida BioClean
- Titanium curettes (Other): Peri-implant pockets will be debrided with titanium curettes.
  Interventions: Other: Titanium curettes

INTERVENTIONS:
Device: Labrida BioClean — The implant pockets will be debrided with the BioClean™ biodegradable brush for 2 minutes and with the brush seated in an oscillating dental handpiece (NSK ESQ10 TEQ) and thereafter irrigated with sterile saline or commercially available and area-specific titanium curettes (Langer and Langer, Rønvig) for 2 minutes and thereafter irrigated with sterile saline. The treatment will be repeated every three months until the terminal examination after 24 months. Debridement is performed with local anaesthesia as needed. Healthy sites will not be retreated.
  Arms: Labrida BioClean
Other: Titanium curettes — Peri-implant pockets will be debrided using titanium curettes.
  Arms: Titanium curettes

SUMMARY:
34 patients diagnosed with mild to moderate peri-implantitis, defined as 2-4 mm peri-implant bone loss, will be randomized to either test treatment with Labrida BioClean® or control treatment with titanium curettes. In total 40 subjects (20 % drop-out rate), treated by 5 clinicians at 5 centers will be included in the study.

DETAILED DESCRIPTION:
4.1 Study design The study will be a prospective multicentre randomized, examiner blinded controlled clinical trial of 24 months duration. Change in mucosal inflammation will be reported after 6 months while the true endpoint parameters i.e., peri-implant attachment will be reported after 1 and 2 years.

4.2 Treatment allocation and blinding Patients will be allocated either to test (Labrida BioClean® or control (titanium curettes) treatment by computer-generated block randomization to ensure equal sample sizes. The examiners will be blinded to the treatment allocation.

4.3 Study setting In total six centres will be included. Patient screening, inclusions and all clinical examinations will be performed by a board-certified specialist in periodontology, registered dental hygienist or specialist in prosthetics at each centre. Treatments will be performed by a dental hygienist or a board-certified specialist in periodontology.

4.4 Patients 40 patients (20+20) diagnosed with mild to moderate peri-implantitis, defined as peri-implant bone loss 2 -4 mm, will be included in the study.

4.5 Recruitment of patients

Patients referred to or seeking care in the included clinics will be screened for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Peri-implantitis defined as 2-4 mm bone loss distally, mesially or both, Probing Pocket Depth (PPD) ≥4mm and inflammation as demonstrated by Bleeding on Probing (mBoP) at least score 2.

In addition to the above mentioned main inclusion criteria, patients can be included if they meet the following conditions:

1. Peri-implantitis as defined above on an implant that has been in function for more than 12 months prior to study start.
2. Above 18 years of age.
3. Eligible for treatment in an outpatient dental clinic (ie, ASA I and II).
4. Had full-mouth plaque scores ≤20% prior to final inclusion and no visual plaque at the included implants prior to study start.
5. Had at least one implant with a loading time of ≥ 12 months prior to baseline.
6. Signed Informed Consent obtained prior to start.
7. Psychological appropriateness.
8. Consent to complete all follow-up visits.

Exclusion Criteria:

Peri-implant bone loss > 4 mm, radiotherapy, chemotherapy, systemic long-term corticosteroid treatment, pregnancy or nursing, anatomical abnormalities, prosthetic factors making access to clinical measurements impossible.

In addition to the above mentioned main exclusion criteria, patients should be excluded if they meet any of the following conditions:

1. Cemented supraconstructions and/or screw retained supraconstructions that for technical reasons makes it impossible to access implant for clinical measurements.
2. Technical complications which according to the examiners judgement has contributed to the disease state and not possible to resolve prior to final inclusion.
3. Mobile implant.
4. Patients diagnosed with periodontal disease must have undergone causative treatment and be re-evaluated.
5. Implants previously treated for peri-implantitis with grafting materials.
6. Receiving medications known to induce mucosal hyperplasia.
7. Uncontrolled diabetes HbA1c > 52, equals 7.0.
8. Receiving systemic antibiotics < 3 months prior to inclusion.
9. Pregnant or lactating.
10. Any condition or current treatment for any condition, which in the opinion of the investigator and/or consulting physician, may constitute an unwarranted risk.
11. Presence of psychological characteristics, such as inappropriate attitude or motivation, which will influence treatment execution and treatment outcome.
12. Unwillingness to undergo treatment.
13. Advanced, untreated and uncontrolled peri-implantitis on neighbouring implants.
14. If, in the opinion of the therapist, conditions are such that dental implants are deemed failing.
15. Ongoing or previous radiotherapy to the head-neck region.
16. Ongoing or previous chemotherapy.
17. Systemic long-term corticosteroid treatment.
18. Patients medicating with warfarine products or similar.

    -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Inflammation | 3 months after first treatment
  Reduction in peri-implant mucositis as measured clinically up to three months after therapy.
Progression of bone loss | 12 months after first treatment.
  True end-point

SECONDARY OUTCOMES:
Morbidity | 3 months
  To compare patient morbidity after use of Labrida BioClean® versus titanium curettes determined on a VAS scale assessed at the 3 month treatment visit.
Adverse events | 12 months
  To assess safety of BioClean™ by evaluating the occurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Caspar Wohlfahrt, PhD, Study Director — Oslo University
Locations (5):
- Norway (3):
  - Spesdent, Oslo
  - Colosseum Majorstuen, Oslo
  - Bjerke Tannmedisin AS, Oslo
- Sweden (2):
  - Odontologiska Institutionen, Jönköping
  - Blekingesjukhuset, Karlskrona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeza B, Wohlfahrt C, Pilloni A. Chitosan brush for professional removal of plaque in mild peri-implantitis. Minerva Stomatol. 2017 Aug;66(4):163-168. doi: 10.23736/S0026-4970.17.04040-7. Epub 2017 May 10. PMID 28497660